CLINICAL TRIAL: NCT06414876
Title: Title: Urinary Oxytocin Levels in Children Receiving Animal-Assisted Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UOLinCRAAT_Uppsala University
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Animal Assisted Therapy
Keywords: Children; Hospital; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The children played with the hospital dog and then by themselves. (Experimental)
  Interventions: Behavioral: Hospital dog
- The children played by themselves and then with the hospital dog. (Experimental)
  Interventions: Behavioral: Hospital dog

INTERVENTIONS:
Behavioral: Hospital dog — The hospital dog always has a well educated dog instructor beside.
  Other Names: The children played with the hospital dog in about 40 minutes.

SUMMARY:
There has been growing interest in animal-assisted therapy (AAT) in recent decades due to increasing reports indicating its health benefits for adult patients. These benefits are partly attributed to changes, usually increased levels of the neuropeptide oxytocin.

Aim: To investigate changes in oxytocin levels in hospitalized children during animal-assisted therapy sessions with a certified hospital dog.

Method: Urine samples were collected from 35 hospitalized children (3-17 years) before and after each participant had a session with the hospital dog. Oxytocin levels were analysed with an acetylcholinesterase (AChE) competitive enzyme-linked immunosorbent assay (ELISA). Creatinine levels were measured to determine the subject's fluid intake and then divided by the hormonal concentration (uOT pg/mg).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized children

Exclusion Criteria:

* Multiresistent bacteria
* Immunosuppressed
* Large burns

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Change in oxytocin levels | Day of enrollment
  Concentration of oxytocin (pg/mg) in urine samples measured by ELISA.

IPD SHARING:
Plan to Share IPD: No